CLINICAL TRIAL: NCT00732446
Title: An Evaluation of the Safety and Efficacy of the Administration of a Fixed Combination of Moxifloxacin 0.5% and Dexamethasone 0.1% Eye Drops Compared With the Individual Administration of Moxifloxacin 0.5% and Dexamethasone 0.1% in the Treatment of Bacterial Ocular Inflammation and Infection (Blepharitis and/or Keratitis and/or Conjunctivitis)
Brief Title: Safety/Efficacy of Antibiotic Steroid Combination in Treatment of Blepharitis and/or Keratitis and/or Conjunctivitis
Acronym: BRA-07-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Rubens Belfort Jr. - Full Professor of Ophthalmology, Federal University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BRA-07-02
Record Dates: First submitted 2008-08-11; First posted 2008-08-12 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2008-08

CONDITIONS: Blepharitis; Conjunctivitis; Keratitis
Keywords: moxifloxacin; dexamethasone; ocular inflammation; ocular infection
MeSH Terms: conditions — Blepharitis; Conjunctivitis; Keratitis; Eye Infections | interventions — Moxifloxacin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): antibiotic /steroid combination compared with individual administration of steroid and antibiotic
  Interventions: Drug: Moxifloxacin; Drug: Dexamethasone
- 1 (Experimental): combination antibiotic steroid compared with individual administration of steroid and antibiotic - new therapeutic indication
  Interventions: Drug: Moxifloxacin and Dexamethasone combined

INTERVENTIONS:
Drug: Moxifloxacin and Dexamethasone combined — moxifloxacin 0,5% qid and dexamethasone 0,1% qid combined
  Other Names: vigadexa
  Arms: 1
Drug: Moxifloxacin — moxifloxacin 0,5% qid and
  Other Names: maxidex and vigamox
  Arms: 2
Drug: Dexamethasone — dexamethasone 0,1% qid
  Arms: 2

SUMMARY:
Safety and efficacy of antibiotic steroid combination compared with individual administration in the treatment of bacterial ocular inflammation and infection (blepharitis and/or keratitis and/or conjunctivitis).

DETAILED DESCRIPTION:
Antibiotic/steroid combination compared to individuals components 8 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of blepharitis and/or keratitis and/or bacterial conjunctivitis

Exclusion Criteria:

* Uncontrolled glaucoma or intraocular hypertension
* Wear contact lens during the study
* Patients with sight in a single eye
* Suspicious of viral, fungic infection
* Use of any other ophthalmic drugs during the study
* Use of immunosuppressant therapy
* Known or suspected allergy or hypersensibility to any component of study medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of ocular sign/symptoms (hyperemia on bulbar conjunctiva, palpebral conjunctiva, conjunctival exsudates, palpebral erythema at final visit (Day 8) | Day 8

SECONDARY OUTCOMES:
Evaluation of sign and symptoms of blepharitis and/or keratitis and/or bacterial conjunctivitis | Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Rubens Belfort, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil